CLINICAL TRIAL: NCT06594380
Title: Observation of Clinical Effect of New Oropharyngeal Airway in Patients With Obstructive Sleep Apnea Hypoapnea Syndrome During Painless Gastroenteroscopy
Brief Title: Observation of Clinical Effect of New Oropharyngeal Airway in Patients With OSHAS During Painless Gastroenteroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianbo Wu (Other)
Responsible Party: Sponsor-Investigator, Jianbo Wu, chief physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2024(084)
Record Dates: First submitted 2024-09-01; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: OSAHS; Gastrointestinal Endoscopy; Airway Complication of Anesthesia
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Using a new oropharyngeal airway set
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Using a new oropharyngeal airway set (Experimental): In the new oropharyngeal airway group (experimental group), oxygen was continuously supplied through a catheter partially attached to the endoscopic bite before induction of anesthesia until the end of gastroenteroscopy
  Interventions: Device: Group using new oropharyngeal airway (experimental group)
- The conventional endoscopic bite group was used (Active Comparator): In the conventional endoscopic bite group (control group), oxygen was continuously supplied through a conventional nasal catheter before induction of anesthesia and until the end of gastroenteroscopy
  Interventions: Device: Endoscopic bite group (control group)

INTERVENTIONS:
Device: Group using new oropharyngeal airway (experimental group) — Before anesthesia induction, study participants in the experimental group received 5-6L/min oxygen for about 1min through an endoscopic bite oxygen supply device, and anesthesia induction was administered with propofol 3mg/kg and sufentanil 7μg.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. When participants achieved sufficient sedation (about BIS40), they were placed into the oropharyngeal airway through the endoscopic bite and began gastroscopy.Anesthetic maintenance was administered with a continuous pump of 5mg/kg·h propofol until completion of the examination
  Arms: Using a new oropharyngeal airway set
Device: Endoscopic bite group (control group) — Prior to induction of anesthesia, control study participants inhaled 5 to 6L/min of oxygen through a nasal catheter for approximately 1 minute.Anesthesia was induced by propofol 3mg/kg and sufentanil 7μg.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. The endoscopic procedure began when the study participants reached sufficient sedation (about BIS40) and the ordinary endoscopic bite group reached sufficient sedation.Anesthetic maintenance was administered with a continuous pump of 5mg/kg·h propofol until completion of the examination.
  Arms: The conventional endoscopic bite group was used

SUMMARY:
the(obstructivesleepapneahypoapneasyndromeOSAHS) is a kind of to sleep appear periodically in the process of syndrome characterized by partial or complete obstruction of upper respiratory tract.Patients with obstruction during the attack, faced with percutaneous arterial blood oxygen saturation (percutaneousarterialoxygensaturation, SpO2) to reduce the risk of can also trigger hypercapnia and cardiovascular dysfunction.The global incidence of OSAS is 4.0% in males and 2.0% in females .Sedative drugs inhibit the response of OSAS patients to external stimuli and may cause pharyngeal muscle collapse, leading to an increased risk of respiratory adverse events during painless gastroscopy in this population .In fact, OSAS has been identified as an independent risk factor for endoscopic hypoxia .Currently, there is no special oropharyngeal ventilation device used during gastroenteroscopy. Recently, a new type of oropharyngeal ventilation channel has been developed and applied in clinic.Compared with the conventional nasal catheter, the new oropharyngeal airway nasal mask can better fit the patient's face, ensure the air tightness inside the nose mask and maximize the oxygen supply efficiency. The carbon dioxide outlet connected to the oropharyngeal airway body can not only collect the patient's exhaled gas, but also reduce the backflow of carbon dioxide gas.It can also access carbon dioxide detection equipment to monitor the patient's PCO2 at the end of breath in real time .In order to evaluate whether the new oropharyngeal airway can reduce the incidence of hypoxia during painless gastroenteroscopy in general patients, the study was designed to investigate the safety and efficacy of the new oropharyngeal airway.

DETAILED DESCRIPTION:
1. The study population was recruited by the principal investigator under strict control, and 130 patients with obstructive sleep apnea hypopnea syndrome (diagnosed as OSAHS by polysomnography monitoring) who underwent painless gastroenteroscopy since the same day were selected. They were informed and agreed to this clinical trial.2. Sample size calculation:According to the pre-test results, the incidence of hypoxia in the test group and the control group were 0.2 and 0.5, respectively. The sample size was calculated using PASS software, and the bilateral test level α=0.05 and the test efficacy power=0.9 were set. 52 cases were required in each group according to the incidence of hypoxia, and 65 cases in each group were calculated after considering 20% shedding rate, totaling 130 cases.3. Specific study contents: Study participants entered the examination room to establish venous access, and used 2% lidocaine gel 5ml containing mouthwash and pharynx.Heart rate (HR), pulse oxygen saturation (SpO2), end-expiratory carbon dioxide, IPI (composite lung index), ECG monitoring, and non-invasive blood pressure (measured every 2.5 minutes) were routinely monitored before anesthesia induction.Ask patient to lie on left side.In this study, the investigators planned to implement simple randomization using SAS: (1) The group using the new oropharyngeal airway (test group) : Oxygen was continuously supplied through a catheter partially attached to the endoscopic mouth before induction of anesthesia until the end of gastroenteroscopy.(2) In the conventional endoscopic bite group (control group), oxygen was continuously supplied through a common nasal catheter before induction of anesthesia until the end of gastroenteroscopy.The entire trial operation process was completed by the investigators participating in the clinical trial.Before induction of anesthesia, study participants in the experimental group received 5-6L/min of oxygen for about 1 minute through an endoscopic biting oxygen supply device, and participants in the control group inhaled 5-6L/min of oxygen for about 1 minute through a nasal catheter.Propofol 3mg/kg and sufentanil 7μg were used to induce anesthesia in both groups.Sufentanil was given at the beginning of pre-oxygen inhalation, and propofol was given 1min later. When participants achieved sufficient sedation (about BIS40), the new oropharyngeal airway group was placed into the oropharyngeal airway through the endoscopic bite and then began gastroscopy.The ordinary endoscopic bite group began to perform endoscopic operation after sufficient sedation was achieved.In both groups, 5mg/kg·h propofol was injected continuously to maintain anesthesia until the examination was completed.If participants showed frowning or slight body movement during diagnosis and treatment, 40 to 50mg of propofol was added intravenously.If HR < 50 times/intravenous injection of atropine 0.5mg;MAP < 60mmHg intravenous hydroxyamine 1mg;When SpO2 < 92%, artificial airway intervention such as jaw support, assisted breathing or mask was given.After the examination, study participants were not allowed to leave the examination room until they had a MOAA/S score of 3-4.If the sedation/anaesthesia Discharge rating scale scores more than 9 points, patients can be accompanied by relatives and friends.The incidence of hypoxia (75%≤SpO2 < 90%, ≤60s) and severe hypoxia (SpO2 < 75% or 75%≤SpO2 < 90%, ≥60s) during anesthesia were recorded.The incidence of choking, reflux aspiration and laryngeal spasm were recorded.The time of intervention was half or disappearance of end-expiratory carbon dioxide and/or disappearance of thoracic fluctuation and/or SpO2 < 95%, that is, opening the airway successively until SpO2≥95%, and recording the last means of opening the airway.The means of opening the airway of the two groups were the same, including: 1) adjusting the oxygen flow;2) Lift the lower jaw;3) Mask ventilation (pull out the gastroscope if necessary);4) Tracheal intubation or laryngeal mask for ventilator assisted ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* evidence of polysleep monitoring for diagnosis of OSAHS
* written informed consent of patient or family member
* painless stomach + colonoscopy
* ASA grade I-II

Exclusion criteria:

* Patients with clotting disorders or a tendency to oropharyngeal bleeding, mucosal damage or space occupation, difficulty in placing oropharyngeal airway, etc., who could not perform oropharyngeal airway ventilation;
* Upper respiratory tract infections such as mouth, nose or throat;
* Fever (core body temperature ≥37.5℃);
* a confirmed diagnosis of pregnancy or breastfeeding;
* Allergic to sedatives such as propofol or equipment such as tape;
* Emergency surgery;
* Multiple trauma;
* SpO2 < 95% before operation;
* A history of drug and/or alcohol abuse within 2 years prior to the start of the screening period;(Drinking more than three times standard alcoholic beverages per day, equivalent to about 10g of alcohol or equivalent to 50g of Chinese liquor);
* Patients with previous psychiatric and neurological diseases, such as depression, severe central nervous depression, Parkinson's disease, basal ganglia disease, schizophrenia, epilepsy, Alzheimer's disease, myasthenia gravis;
* Currently participating in other clinical trials;
* Patients who are deemed unfit by the investigator to participate in the trial;
* Patients with a history of smoking should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxia | 1 minute after anesthesia induction
  The incidence of hypoxia (75% ≤ SpO2 < 90%, ≤ 60s)

SECONDARY OUTCOMES:
The incidence of severe hypoxia | 1 minute after anesthesia induction
  The incidence of severe hypoxia (SpO2 < 75% or 75% ≤SpO2 < 90%, ≥60s)
The incidence of requiring airway intervention | 1 minute after anesthesia induction
  Tracheal intubation and noninvasive ventilation are required
The dosage of additional drugs was recorded during the operation | 1 minute after anesthesia induction
  The dosage of additional drugs was recorded during the operation
The satisfaction of endoscopists was recorded | Within 30 minutes after anesthesia awakening
  Patient satisfaction scales usually use a 0-10 scale, where 0 is very dissatisfied and 10 is very satisfied.Patients are asked to select a number on the rating scale to indicate satisfaction with medical services or pain relief methods based on their actual experience
Recorded adverse events | 1 minute after anesthesia induction
  The incidence of choking, laryngeal spasm and reflux aspiration were observed.Apnea or slow breathing episodes (defined as respiratory rate ≤6 beats/min);Bradycardia is defined as a heart rate ≤50 beats/min.Serious adverse events such as tracheal intubation, non-invasive ventilation, use of vasopressors, and hospitalization are required.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Wu, Principal Investigator — Shandong First Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] You Q, Liu X, Meng Y, Zhu Y, Sun C, Wu J. Clinical effects of the use of a novel oropharyngeal airway in painless gastroscopy in patients with obstructive sleep apnoea-hypopnoea syndrome: a randomised controlled trial protocol. BMJ Open. 2026 Jan 27;16(1):e094885. doi: 10.1136/bmjopen-2024-094885. PMID 41592820

DOCUMENTS (1):
  • Study Protocol (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT06594380/Prot_000.pdf